CLINICAL TRIAL: NCT04830917
Title: Prospective Randomized Clinical Trial Comparing Kinesiotape and Oval 8 to Quick Cast for Conservative Treatment of Mallet Finger Injury
Brief Title: Conservative Treatment of Mallet Finger Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Specialty Group PC, Fairfield (Other)
Responsible Party: Principal Investigator, Lori Algar, Hand therapist/occupational therapist, Orthopaedic Specialty Group PC, Fairfield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVMC 17-328
Record Dates: First submitted 2021-03-30; First posted 2021-04-05 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Conservatively Treated Mallet Finger Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with Kinesiotape and Oval 8 (Experimental)
  Interventions: Other: Immobilization type for mallet injury
- Treatment with quick cast (Experimental)
  Interventions: Other: Immobilization type for mallet injury

INTERVENTIONS:
Other: Immobilization type for mallet injury — Method to hold the DIP joint in full extension to allow healing of terminal tendon injury/mallet injury

SUMMARY:
Comparing outcomes of individuals treated with Kinesiotape and oval 8 versus quick cast for a conservatively managed mallet finger injury. Outcomes include DIP joint extension lag, patient satisfaction and function via the MHQ.

ELIGIBILITY:
Inclusion Criteria:

* determined by a physician to require conservative treatment for a mallet finger injury, at least 18 years of age

Exclusion Criteria:

* previous injury to the involved digit impacting ROM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Goniometric measurement of range of motion for distal interphalangeal joint extension lag at the involved digit | 12 weeks from injury

SECONDARY OUTCOMES:
Goniometric measurement of range of motion for distal interphalangeal joint extension lag at the involved digit | 6 months post injury
Brief Michigan Hand Outcome Questionnaire | 12 weeks from injury
Brief Michigan Hand Outcome Questionnaire | 6 months post injury
Satisfaction on a visual analog scale (0-10) | 12 weeks from injury
Satisfaction on a visual analog scale (0-10) | 6 months post injury
Goniometric measurement of range of motion deficit for distal interphalangeal joint flexion for involved digit | 12 week post injury
Goniometric measurement of range of motion deficit for distal interphalangeal joint flexion for involved digit | 6 months post injury
Pain according to a numeric pain rating scale (0-10/10) | 12 weeks after injury
Pain according to a numeric pain rating scale (0-10/10) | 6 months post injury

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Specialty Group PC, Fairfield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided